CLINICAL TRIAL: NCT02499692
Title: SYNERGY China: A Prospective, Multicenter Trial to Assess the SYNERGYTM MONORAILTM Everolimus-Eluting Platinum Chromium Coronary Stent System for the Treatment of Atherosclerotic Lesion(s)
Brief Title: SYNERGY China: Assess SYNERGY Stent in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2342
Record Dates: First submitted 2015-04-30; First posted 2015-07-16 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYNERGYTM Coronary Stent System (Experimental): Device:SYNERGY MONORAIL Everolimus-Eluting Platinum Chromium Coronary Stent System
  Interventions: Device: SYNERGYTM Coronary Stent System

INTERVENTIONS:
Device: SYNERGYTM Coronary Stent System — SYNERGYTM MONORAILTM Everolimus-Eluting Platinum Chromium Coronary Stent System

SUMMARY:
Prospective, multicenter, single-arm study, enroll 100 patients in no more than 10 sites across China, the primary endpoint is Technical success.

DETAILED DESCRIPTION:
The study is To evaluate clinical and peri-procedural angiographic outcomes for the SYNERGYTM MONORAILTM Everolimus-Eluting Platinum Chromium Coronary Stent System in the treatment of subjects with atherosclerotic lesion(s) ≤34 mm in length (by visual estimate) in native coronary arteries ≥2.25 mm to ≤4.0 mm in diameter (by visual estimate).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject must be at least 18 -75 years of age
2. Subject is eligible for percutaneous coronary intervention (PCI)
3. Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.25 mm and ≤4.0 mm, length must be ≤34* mm (by visual estimate), Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1

Key Exclusion Criteria:

1. Planned PCI (including staged procedures) or CABG after the index procedure
2. Subject with out of range complete blood count (CBC) values that are determined by the study physician to be clinically significant.
3. Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
4. Planned treatment of more than 3 lesions, Planned treatment of lesions in more than 2 major epicardial vessels, Planned treatment of a single lesion with more than 1 stent
5. Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate.
6. Target vessel develops a dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C following the pre-dilatation/pre-treatment of the first target lesion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yalin Han, Principal Investigator — Shenyang Northern Hospital (The General Hospital of Shenyang Military Region)
Locations (8):
- China (8):
  - AeroSpace center hospital, Beijing
  - the second hospital of Jilin Unversity, Changcun
  - Daqing General Oil Field Hospital, Daqing
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - The First Hospital of Lanzhou University, Lanzhou
  - General Hospital of SY Military Institute, Shenyang
  - TEDA International Cardiovascular Hospital, Tianjin
  - Wuhan Asia Heart Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SYNERGYTM Coronary Stent System
Started | 103
Completed | 103
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.92 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Technical Success Rate
Description: Technical success rate, defined as successful delivery and deployment of the study stent to the target lesion, without balloon rupture or stent embolization, and post-procedure diameter stenosis of <30% assessed in 2 near-orthogonal projections with TIMI 3 flow in the target lesion, as visually assessed by the physician
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
percentage of participants | 98.1

2. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
percentage of participants | 0

3. Secondary Outcome: Target Lesion Failure (TLF) Rate
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
percentage of participants | 0

4. Secondary Outcome: Target Vessel Revascularization (TVR) Rate
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
percentage of participants | 0

5. Secondary Outcome: Target Vessel Failure (TVF) Rate
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
percentage of participants | 0

6. Secondary Outcome: Myocardial Infarction (MI, Q-wave and Non-Q-wave) Rate
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | SYNERGYTM Coronary Stent System
Number analyzed (Participants) | 103
percentage of participants | 0

ADVERSE EVENTS:
Arm/Group | SYNERGYTM Coronary Stent System
Serious Adverse Events (participants affected / at risk) | 1/103
Other Adverse Events (participants affected / at risk) | 7/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGYTM Coronary Stent System (N=103)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNERGYTM Coronary Stent System (N=103)
Cardiac disorders (Cardiac disorders) | 2 (2)
General disorders and administration site conditions (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less